CLINICAL TRIAL: NCT05556070
Title: Brighter Bites & University of Texas Physicians Produce Rx: Evaluating the Effectiveness of a Prospective Clinical Nutrition Study With Produce Prescriptions
Brief Title: Brighter Bites & UT Physicians Produce Rx Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Brighter Bites (Unknown)
Responsible Party: Principal Investigator, Christine Markham, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-22-0629
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Other: Arm 1; Other: Brighter Bites app
- Arm 2 (Experimental)
  Interventions: Other: Arm 2; Other: Brighter Bites app
- Arm 3 (Active Comparator)
  Interventions: Other: Arm 3

INTERVENTIONS:
Other: Arm 1 — : Local retailer produce vouchers ($25 value) will be distributed to the families biweekly over a 32-week period for a total of 16 vouchers. The vouchers can be redeemed for fresh produce at the grocery store that issued the vouchers.
  Arms: Arm 1
Other: Arm 2 — Boxes of fresh fruits and vegetables (F&V), each containing approximately 50 servings of F&V, will be assembled by Brighter Bites at school sites using donated produce and delivered to houses using DoorDash. F&V boxes will be distributed to families every 2 weeks over 32 weeks.
  Arms: Arm 2
Other: Arm 3 — subjects in this arm will receive the usual standard of care at the clinic for the study period
  Arms: Arm 3
Other: Brighter Bites app — Participants in Arms 1 and 2 will also receive nutrition education using the Brighter Bites app which includes recipes for a variety of meal types or produce types, all of which are searchable. Recipes include the average cost to prepare, the number of servings, and the calories for the recipe. The Brighter Bites app also includes healthy living "Brighter Choices" suggestions such as tips for how to store different types of foods, gardening tips, and tips to pack a healthy lunchbox. In addition to the Brighter Bites app, trained staff will facilitate virtual nutrition education for patient families.
  Arms: Arm 1; Arm 2

SUMMARY:
The purpose of this study is to clinically evaluate the effectiveness of an at-home produce delivery prescription or grocery store vouchers prescription at improving weight status and obesity-related health outcomes of participants across the two clinics as compared to a control group and to examine the impacts of the program on child dietary behavioral outcomes (child fruit and vegetable intake, junk food consumption, and eating at any type of restaurant), and parent feeding practices (preparing foods from scratch, use of nutrition facts labels to make purchasing decisions, and eating meals with their referent child)

ELIGIBILITY:
Inclusion Criteria:

* reside within a 10-mile radius of a Brighter Bites school
* Medicaid recipients or low-income uninsured
* parents must be able to read and write in English or Spanish to complete surveys

Exclusion Criteria:

* currently participating in Brighter Bites
* with a family member/sibling currently participating in Brighter Bites
* child is currently attending a school that offers Brighter Bites

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline, 9 months after baseline
Change in systolic blood pressure | Baseline, 9 months after baseline
Change in diastolic blood pressure | Baseline, 9 months after baseline
Change in hemoglobin A1c | Baseline, 9 months after baseline
Change in Aspartate transaminase (AST) | Baseline, 9 months after baseline
Change in alanine aminotransferase (ALT) | Baseline, 9 months after baseline
Change in Lipid panel | Baseline, 9 months after baseline

SECONDARY OUTCOMES:
Change in amount of fruit and vegetable intake | Baseline, 9 months after baseline
Change in amount of junk food consumed | Baseline, 9 months after baseline
Change in number of times subject eats out at restaurants | Baseline, 9 months after baseline
Change in parent feeding practices as assessed by the number of times parent has cooked food from scratch | Baseline, 9 months after baseline
Change in parent feeding practices as assessed by the number of times parent has used nutrition facts labels to make purchasing decisions | Baseline, 9 months after baseline
Change in parent feeding practices as assessed by the number of times parent has eaten meals with their referent child | Baseline, 9 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christine Markham, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No